CLINICAL TRIAL: NCT06154863
Title: Evaluation of Recurrence in Patients With Differentiated Thyroid Cancer
Brief Title: Recurrence in Patients With Differentiated Thyroid Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Salah Mahmoud, Principal Investigator, Assiut University
Other Study IDs: recurrence in thyroid cancer
Record Dates: First submitted 2023-11-22; First posted 2023-12-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Differentiated Thyroid Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: RAI — Radioactive iodine

SUMMARY:
The aim of this study is to assess the recurrence-free survival (RFS) rate and recurrence-related factors, especially the relationship between RFS and RAI dose, in patients who received RAI after thyroidectomy.

DETAILED DESCRIPTION:
Thyroid cancer is the most frequent cancer of the endocrine system, and its incidence is constantly rising worldwide. This is mainly because of advances in examination modalities that have made it possible to detect smaller cancers at an early stage.

Owing to advancements in screening techniques and treatment methods, the number of patients who die from thyroid cancer is small compared to the incidence.[1]

The most common type of thyroid cancer is differentiated thyroid cancer (DTC), which includes papillary and follicular carcinomas. Women are three times more likely to develop thyroid cancer than men. [2] Adjuvant RAI131 (AT) is recommended post thyroidectomy, because of its therapeutic impact on micro-invasions or micro-metastases, to reduce the likelihood of recurrence in patients who do not have metastases but have risk of recurrence according to the Japanese guidelines and American Thyroid Association guidelines [3],[4].

AT could prolong the survival of patients with intermediate-risk DTC [5]. Additionally, a meta-analysis has shown that AT is effective in reducing recurrence in some studies but not in others, and the effect of AT on recurrence prevention, especially in high-risk DTC, remains unclear.[6].

Although there are reliable reports discussing the relationship between the success or failure of remnant ablation [7],[8], recurrence after AT is rarely reported and the number of cases is small. In addition, no study has so far discussed the relationship between the success or failure of AT or remnant ablation and recurrence or death [9],[10].

ELIGIBILITY:
Inclusion Criteria:

* Patients with DTC (differentiated thyroid cancer) who underwent total or subtotal thyroidectomy without distant metastasis and gross residual tumors.
* Followed by ablation with RAI and underwent post RAI whole body scan.
* Having baseline TG (thyroglobulin), Anti-TG antibodies (anti thyroglobulin) and neck US.
* Patients with lymph node metastasis will be included if their lymph nodes had been dissected and no unresectable disease remained.

Exclusion Criteria:

* Patients who received RAI and missed follow-up.
* Patients with no surgical or pathological data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with differentiated thyroid cancer underwent total thyroidectomy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of recurrence-free survival after RAI therapy in patients with thyroid cancer. | 2 years
  Assessment of recurrence-free survival after radioactive iodine-131 therapy in patients with differentiated thyroid carcinoma.

SECONDARY OUTCOMES:
Correlation analysis of I-131 SPECT/CT uptake parameters with the success ablation treatment of thyroid remnant. | 2 years
  Correlation analysis of I-131 SPECT/CT uptake parameters with the success ablation treatment of thyroid remnant in patients with low-intermediate-risk differentiated thyroid cancer.

OTHER OUTCOMES:
Assessment of Prognostic significance of pathological data post thyroidectomy in thyroid cancer. | 2 years
  Assessment of Prognostic significance of pathological data post thyroidectomy in patients with differentiated thyroid cancer.
Assessment of Prognostic significance of anti-thyroglobulin level in differentiated thyroid cancer. | 2 years
  Assessment of Prognostic significance of anti-thyroglobulin level in follow up of patients with differentiated thyroid cancer patients.
Assessment of Prognostic significance of thyroglobulin level in differentiated thyroid cancer. | 2 years
  Assessment of Prognostic significance of thyroglobulin level in follow up of patients with differentiated thyroid cancer.

REFERENCES:
- [Background] Vigneri R, Malandrino P, Vigneri P. The changing epidemiology of thyroid cancer: why is incidence increasing? Curr Opin Oncol. 2015 Jan;27(1):1-7. doi: 10.1097/CCO.0000000000000148. PMID 25310641
- [Background] Sawka AM, Carty SE, Haugen BR, Hennessey JV, Kopp PA, Pearce EN, Sosa JA, Tufano RP, Jonklaas J. American Thyroid Association Guidelines and Statements: Past, Present, and Future. Thyroid. 2018 Jun;28(6):692-706. doi: 10.1089/thy.2018.0070. Epub 2018 Apr 26. PMID 29698130
- [Background] Ruel E, Thomas S, Dinan M, Perkins JM, Roman SA, Sosa JA. Adjuvant radioactive iodine therapy is associated with improved survival for patients with intermediate-risk papillary thyroid cancer. J Clin Endocrinol Metab. 2015 Apr;100(4):1529-36. doi: 10.1210/jc.2014-4332. Epub 2015 Feb 2. PMID 25642591
- [Background] Jeong SY, Lee SW, Kim WW, Jung JH, Lee WK, Ahn BC, Lee J. Clinical outcomes of patients with T4 or N1b well-differentiated thyroid cancer after different strategies of adjuvant radioiodine therapy. Sci Rep. 2019 Apr 3;9(1):5570. doi: 10.1038/s41598-019-42083-3. PMID 30944403
- [Background] Lee SH, Roh JL, Gong G, Cho KJ, Choi SH, Nam SY, Kim SY. Risk Factors for Recurrence After Treatment of N1b Papillary Thyroid Carcinoma. Ann Surg. 2019 May;269(5):966-971. doi: 10.1097/SLA.0000000000002710. PMID 29462007